CLINICAL TRIAL: NCT03349047
Title: Trial To Reduce Food Allergy Anxiety by Holding the Allergen (TOUCH Study)
Brief Title: Anxiety About Casual Exposure to Food Allergens
Acronym: TOUCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-1957
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Food Allergy
Keywords: Food Allergy; Anxiety; Casual Exposure; Peanut Hypersensitivity; Tree nut Hypersensitivity; Adolescents
MeSH Terms: conditions — Food Hypersensitivity; Anxiety Disorders; Peanut Hypersensitivity; Nut Hypersensitivity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Active Comparator): Behavioral Intervention Group - Education regarding nut allergy and will also have contact with nut.
  Interventions: Behavioral: Behavioral intervention group; Behavioral: Education
- Control (Placebo Comparator): Education regarding nut allergy
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Behavioral intervention group — Patients will hold the peanut or tree nut in a cup and will be asked to touch the nut with their finger.
  Arms: Behavioral Intervention
Behavioral: Education — The group will be educated about what can occur with contact with or being in proximity of peanuts or tree nuts.

SUMMARY:
Living with food allergy may result in anxiety and reduced quality of life. Food allergic patients and their families are often concerned about casual exposure with the offending allergen through skin contact or being near the offending food, which is actually very low risk. This concern can limit social activities and increase stress. The aim of this study is to provide a behavioral intervention consisting of having peanut/tree nut allergic patients hold a cup with a peanut or tree nut to which the patient is allergic to and touching it. The goal is to reduce anxiety about casual exposure to food allergens and improve quality of life for patients with food allergies and their families.

DETAILED DESCRIPTION:
The purpose of the present study is to determine if having patients (ages 9-17) who are peanut and/or tree nut allergic, and endorse anxiety/discomfort about non-ingestion exposure, hold and touch their offending allergen in addition to education leads to reduced discomfort for both patient and caregiver compared to education alone. The primary outcome measure is immediate differences in the score obtained on a child-reported scale in response to a question assessing how worried the patient is about the thought of being near or touching peanut or tree nut from pre-intervention to immediate post-intervention when compared between an intervention (education and touching) and a control group (education only). Secondary outcome measures include: difference between and within groups of child-reported scales regarding questions assessing patients worry regarding casual exposure immediately and one month post intervention within and between groups, differences between and within groups on a parent-reported scale regarding parental worry about casual exposure to food allergen immediately and one month post intervention within and between groups, differences between and within groups on a parent-proxy measures regarding child worry about casual exposure to food allergen immediately and one month post intervention within and between groups, improvement in child anxiety and parent-proxy measures of anxiety from pre-intervention to one month post-intervention within and between groups and improvement in parent-proxy measures of quality of life from pre-intervention to one month post-intervention within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 9 years to 17.5 years
* Patient seen in the outpatient clinic (no inpatients).
* Patient and or caretaker endorses anxiety about being in proximity with or touching peanut
* Patients must have been diagnosed with a peanut and or tree nut allergy

Exclusion Criteria:

* Patients and caregiver(s) without ability to understand the study, as determined by either: a previously diagnosed cognitive disability or inability to repeat the study protocol at the time of consent.

Ages: 108 Months to 210 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Child worry about casual exposure | Baseline and approximately 10 minutes
  Change in a child-reported 10-point likert scale assessing how worried the child is about the thought of being near or touching peanut or tree nut, where 0 is not worried at all and 10 is extremely worried pre-intervention compared to immediately post-intervention.

SECONDARY OUTCOMES:
Parent worry about casual exposure | Baseline and one month
  Parent-proxy reported scale in response to additional questions assessing how worried the child is about the thought of being near or touching peanut or tree nut, where 0 is not worried at all and 10 is extremely worried, at one month compared to baseline.
Food Allergy Quality of Life-Parental Burden (FAQL-PB) Questionnaire | One month
  The score obtained on a parent-reported quality of life questionnaire (QOL). QOL is measured on a standardized FAQL-PB questionnaire which consists of 17 questions and responses are measured on a 6-point likert scale where 0 is not limited and 6 is very limited with total from 0 to 102.
The Screen for Child Anxiety Related Disorders (SCARED) | Baseline and one month
  Change in child anxiety at one month compared to baseline.The SCARED consists of 17 items, rated on a 3 point Likert-type scale. Total score range from 0 (not anxious) to 34 (very anxious).
SCARED - parent version | Baseline and one month
  Change in parent-proxy measures of child anxiety on parent reported SCARED at one month compared to baseline. 17 items, rated on a 3 point Likert-type scale. Total score range from 0 (not anxious) to 34 (very anxious).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sicherer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No